CLINICAL TRIAL: NCT06696846
Title: Cord Blood-derived CD70-targeting CAR-NK Cell Therapy for Refractory/relapsed T Cell Lymphoma and Acute Myeloid Leukemia
Brief Title: CD70-CAR-NK Cell Therapy for T Cell Lymphoma and Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0992
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Relapsed/refractory T-cell Lymphoma; Relapsed/refractory Acute Myeloid Leukemia
Keywords: CD70; CAR-NK; T cell lymphoma; acute myeloid leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD70 CAR-NK for the treatment of CD70-positive relapsed/refractory T-cell lymphoma and AML (Experimental): The first stage is a dose escalation study, with three CD70 CAR-NK dose levels. Each dose level is planned to recruit 3 to 6 subjects to evaluate safety and efficacy and determine the number of CD70 CAR-NK cells for treatment in the second stage. The second stage is the dose expansion stage, where 30 subjects are recruited to receive the number of CD70 CAR-NK cells recommended in the first stage.
  Interventions: Biological: CD70 CAR-NK

INTERVENTIONS:
Biological: CD70 CAR-NK — CAR - NK cells constructed by using genetic engineering technology retain the original extensive tumor - killing ability of NK cells. By using their unique target cell recognition mechanism, the target is accurately locked on specific antigen proteins, thereby enhancing the anti - tumor effect. Cord blood-derived CAR - NK cell products shorten the treatment time and are inexpensive. Multiple studies have confirmed the feasibility of CAR - NK cells in treating hematological tumors.
  Blocking the CD70/CD27 signaling pathway plays an important role in inhibiting CD70 - positive tumors, such as refractory/relapsed T - cell lymphoma and acute myeloid leukemia. Pre - clinical studies in our laboratory have proved that CD70 CAR - NK can effectively inhibit the in - vivo and in - vitro proliferation of T - cell lymphoma and prolong survival.

SUMMARY:
CD70 is a promising target for immunotherapy because it is overexpressed in T-cell lymphoma (TCL) and acute myeloid leukemia (AML) tumor cells but is found in deficient levels in normal tissues and hematopoietic stem cells. This study aims to evaluate the safety and efficacy of CD70-targeted CAR-NK (CD70-CAR-NK) cells in patients with relapsed and refractory TCL and AML.

DETAILED DESCRIPTION:
Despite significant advances in CAR-T cell therapy for refractory and relapsed B-cell malignancies and multiple myeloma, CAR-T therapy for T cell lymphoma and acute myeloid leukemia only resulted in suboptimal response partly due to the lack of an ideal target and possible fratricide. Chimeric antigen receptor (CAR)-NK cells may have advantages over CAR-T cells, such as reducing cytokine release and preventing fratricide and tumor contamination in T-cell lymphoma. CD70, which is overexpressed in tumor cells in T cell lymphoma and AML but minimally in normal tissues or hematopoietic stem cells, has emerged as a novel immunotherapy target. Inhibition of the growth of CD70-positive tumors through blocking the CD70/CD27 pathway potentially led to clinical response in relapsed/refractory T-cell lymphoma and AML.

In preclinical studies, we and others have shown that CD70 CAR-NK cells effectively suppress the growth of lymphoma and AML xenograft in vivo, extending the survival of tumor-bearing mice but without significant toxicities. This study aims to evaluate the safety, pharmacokinetics, and efficacy of CD70-targeted CAR-NK cells in patients with CD70-positive relapsed/refractory T-cell lymphoma and AML.

ELIGIBILITY:
Inclusion Criteria:

According to the WHO disease classification, patients with relapsed/refractory T - lymphoma and acute myeloid leukemia:

1. Voluntarily participate in this study and sign the informed consent form;
2. Aged between 18-75 years old, both male and female are eligible;
3. Relapsed/refractory T cell lymphoma is defined as: relapsed/refractory after having received at least two or more lines of previous treatment (patients with anaplastic large -cell lymphoma must have been exposed and resistant to Brentuximab vedotin). The celluar subtypes of T-cell lymphoma include: angioimmunoblastic T-cell lymphoma; peripheral T - cell lymphoma not otherwise specified; ALK-negative anaplastic large - cell lymphoma; Relapsed/refractory AML is defined as: leukemia cells reappear in the peripheral blood after complete remission or the blasts in the bone marrow ≥ 5% or the extramedullary leukemia infiltration outside. Or newly diagnosed cases did not achieve a CR after two courses of standard regimens; those who relapse within 12 months after CR after consolidation and intensification treatment; those who relapse after 12 months and have not responded to conventional chemotherapy; those who relapse two or more times; those with persistent extramedullary leukemia;
4. The expected survival period ≥ 12 weeks;
5. CD70 expression is positive in tumor tissue puncture sections/tumor cells detected by flow cytometry, and the number of CD70 - positive cells detected by immunohistochemistry ≥ 20% (++ or more);
6. ECOG score is 0 - 2;
7. Adequate organ function reserve:

   * Alanine aminotransferase and aspartate aminotransferase ≤ 2.5× UNL;
   * Creatinine clearance rate (Cockcroft - Gault method) ≥ 60 mL/min;
   * Serum total bilirubin and alkaline phosphatase ≤ 1.5× UNL;
   * Glomerular filtration rate > 50 ml/min;
   * Cardiac ejection fraction ≥ 45%;
   * Under indoor natural air environment, the basic oxygen saturation > 92%;
   * Routine blood test: absolute neutrophil count > 1000/mm3, platelet count ≥ 45×109, hemoglobin ≥ 8.0g/dl (the standard for AML patients is ≥ 7.0g/dl; blood transfusion is allowed);
8. Previous autologous hematopoietic stem cell transplantation is allowed once;
9. Patients who have previously received CAR - T cell therapy and were evaluated as ineffective after 3 months or relapsed after CR are allowed;
10. Female subjects of childbearing age must have a negative pregnancy test and agree to take effective contraceptive measures during the trial period;
11. No active lung infection, and indoor air blood oxygen saturation ≥ 92%;
12. Before the study drug is used, approved anti - tumor treatment methods, such as systemic chemotherapy, whole - body radiotherapy, and immunotherapy, have been completed for at least 3 weeks; the wash - out period for targeted drug regimens without chemotherapy is 2 weeks;
13. Two negative tests for COVID - 19 or influenza A.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible for this study:

1. Those with a history of allergy to any component in the cellular product;
2. Those with a history of other tumors;
3. Those who had grade II - IV (Glucksberg criteria) acute GvHD or extensive chronic GvHD after previous allogeneic hematopoietic stem cell transplantation; or those who are currently receiving anti - GvHD treatment;
4. Those who have received gene therapy within the past 3 months;
5. Those with active infections requiring treatment (except for simple urinary tract infections and bacterial pharyngitis). However, prophylactic antibiotic, antiviral, and antifungal treatments are permitted;
6. Subjects with hepatitis B (HBsAg - positive, but HBV - DNA < 103 is not an exclusion criterion) or hepatitis C virus infection (including virus carriers), syphilis, and other acquired or congenital immunodeficiency diseases, including but not limited to those infected with the AIDS virus;
7. Subjects with grade III or IV cardiac insufficiency according to the New York Heart Association cardiac function classification standard of the United States;
8. Those whose toxic reactions from previous anti - tumor treatment have not recovered (CTCAE 5.0 toxic reactions have not recovered to ≤ grade 1, except for fatigue, anorexia, and alopecia);
9. Subjects with a history of epilepsy or other central nervous system diseases;
10. Lactating women who are unwilling to stop breastfeeding;
11. Any other circumstances that, in the opinion of the investigator, may increase the risk to the subject or interfere with the test results;
12. Those with positive nucleic acid tests for COVID - 19 or influenza A.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and type of dose-limiting toxicity (DLT) within 28 days | 28 days
  To determine the incidence and type of dose-limiting toxicity (DLT) within 28 days after CD70-CAR - NK cell infusion
the incidence and severity of treatment-related adverse events as assessed by CTCAE v4.0 | within 90 days after CAR-NK infusion
  CAR-NK treatment-related AEs include CRS, ICANS, cytopenia, and other non-hematological toxicities

SECONDARY OUTCOMES:
Objective response rate (ORR) at day 30 | 30 days
  To evaluate the overall response rate (PR+CR )as assessed by PET-CT for T cell lymphoma, and by bone marrow examination for AML
duration of response | 2 years
  duration of response measured as the time from the date of first documentation of response to the date of first documented progression
progression-free survival | 2 years
  defined as the time from the date of randomization to the date of first documentation of disease progression based on NCCN criteria as evaluated by an independent review committee (IRC), or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
CAR copies as assessed by qPCR | 6 months
  CAR copies in peripheral blood will be monitored by qPCR within 6 months
phenotypes of CAR-NK cells as assessed by flow cytometry | 1 year
  the proportions of CAN-NK cells with different immunophenotypes

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol